CLINICAL TRIAL: NCT04463732
Title: The Relationship Between Maximal Oxygen Consumption and Inspiratory Muscle Activation Pattern Under Loaded Inspiratory Muscle Tests in Healthy Adults
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202005050RINA
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-06

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy group: Subjects are above 20 years old. Their condition is healthy with no history of inspiratory disease. They can cooperate with the measurements of this study.
  Interventions: Other: Loaded inspiratory muscle test and cardiopulmonary exercise test

INTERVENTIONS:
Other: Loaded inspiratory muscle test and cardiopulmonary exercise test — This is an observational study. Loaded inspiratory muscle test is setting at 30% of maximal inspiratory pressure. Subjects will perform only 15 breaths under this intensity to exam the performance of their inspiratory muscles. Loaded inspiratory muscle test is not for training. Cardiopulmonary exercise test is performed by using bicycle ergometer. These two tests will be performed at least 1 week separately.

SUMMARY:
Maximal oxygen consumption, VO2max, is the gold standard to evaluate human aerobic fitness, which stands for the maximal capacity of cardiorespiratory system and musculoskeletal system to transport and utilize oxygen. Previous study showed that there is significant correlation between maximal oxygen consumption from cardiopulmonary exercise test and strength and endurance of lower extremities. In people with sedentary lifestyle, they often limited by the lower limb muscle performance during cardiopulmonary exercise test. Their breathing patterns are more irregular than athletes during cardiopulmonary exercise test. However, there is no study comparing the activation pattern of respiratory muscles between these two groups. Whether the breathing pattern in people with lower exercise capacity is less efficient under exertional activities still unknown. The purpose of this study is to investigate the relationship between maximal oxygen consumption and inspiratory muscle activation pattern in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (age > 20 years old)
* Be able to cooperate with the measurements of this study

Exclusion Criteria:

* any clinical diagnosis that will influence the measurement, including any history of neuromyopathy
* angina, acute myocardial infarction in the previous one month
* pregnancy
* history of syncope during exercise
* any musculoskeletal system disorder that unable to perform cardiopulmonary exercise test

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy population is free from abnormal breathing pattern caused by disease. Their terminals of cardiopulmonary exercise test are not limited by symptoms of disease.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Diaphragm and Sternocleidomastoid muscle activation | during the loaded inspiratory muscle test condition; it would take about 3 minutes
  Root mean square values
Maximal exercise capacity | during the cardiopulmonary exercise test; it would take about 12 to 15 minutes
  Maximal oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, PhD, Study Chair — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy of National Taiwan University, Taipei, Zhongzheng Dist, Taiwan